CLINICAL TRIAL: NCT00001532
Title: Role of Genetic Factors in the Pathogenesis of Lung Disease
Brief Title: Role of Genetic Factors in the Development of Lung Disease
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Suburban Hospital (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960100; 96-H-0100
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01-08

CONDITIONS: Cystic Fibrosis; Pulmonary Fibrosis; Tuberous Sclerosis; Asthma; Pulmonary Sarcoidosis
Keywords: Genetic Polymorphism; Nitric Oxide Synthesis; Alpha 1-Antitrypsin; Candidate Genes; Lung Pathology; Natural History; Lung Disease; Cystic Fibrosis; Asthma
MeSH Terms: conditions — Cystic Fibrosis; Pulmonary Fibrosis; Tuberous Sclerosis; Asthma; Sarcoidosis, Pulmonary; alpha 1-Antitrypsin Deficiency; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Subjects with pulmonary disease or possible pulmonary disease and Relatives
- 2: Healthy

SUMMARY:
This study is designed to evaluate the genetics involved in the development of lung disease by surveying genes involved in the process of breathing and examining the genes in lung cells of patients with lung disease.

The study will focus on defining the distribution of abnormal genes responsible for processes directly involved in different diseases affecting the lungs of patients and healthy volunteers.

Optional CT Sub-study

The standard CT scan will be compared to the low dose radiation CT scan for the 150 subjects enrolled in the sub-study to assess the variation between the two techniques. Specifically, the quantitative computer aided detection of lung CT abnormalities from LAM can be compared to assess whether low radiation dose CT exams is an alternative to conventional CT to monitor disease

status.

This optional sub-study will be offered to up to 100 adult subjects with lung disease and up to 50 children age 9 and older with CF. Children will not be enrolled in the optional CT sub-study unless they have had a standard CT scan for medical purposes to use in comparison. One additional low dose radiation CT scan of the chest may be done as part of this sub-study when these subjects have their next annual CT scan.

DETAILED DESCRIPTION:
This study is designed to evaluate genetic mechanisms of lung disease by surveying polymorphic genes involved in respiratory function and examining gene expression in the lung cells of individuals with pulmonary disease (e.g., alpha 1-antitrypsin deficiency, asthma, chronic obstructive pulmonary disease, cystic fibrosis, sarcoidosis, history of infection, and genetic mutations consistent with lung pathology). Emphasis will be on defining the distribution of allelic variants of nitric oxide synthase, alpha 1-antitrypsin, and the cystic fibrosis transmembrane conductance regulator genes in patients and in age- and sex-matched healthy individuals in a control population.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for patients with AAT deficiency include: (1) Diagnosis of AAT with a confirmed phenotype considered in the high risk category; (2) Clinical phenotype consistent with potential genetic diseases and other genetic causes of lung diseases (3) symptoms consistent with pulmonary disease; (4) chest x-ray consistent with pulmonary disease; (5) pulmonary function tests consistent with pulmonary disease; (6) smokers, defined as individuals who are current smokers (1 pack per day for at least 2 years) and nonsmokers, defined as never-smokers or ex-smokers who have quit smoking three or more years ago;

Inclusion criteria for individuals with chronic obstructive pulmonary diseases include:

1. symptoms consistent with pulmonary disease
2. chest x-ray consistent with pulmonary disease
3. pulmonary function tests consistent with pulmonary disease;
4. smokers, defined as individuals who are current smokers (1 pack per day for at least 2 years) and nonsmokers, defined as never-smokers or ex-smokers who have not smoked for three or more years.

Inclusion criteria for patients with cystic fibrosis include a defined genetic mutation (i.e., any of the known variants of the CFTR gene, such as delta F508 allele) or a cystic fibrosis phenotype and clinical features consistent with this disease. Children with cystic fibrosis over eight years of age may be included.

Patients with established diagnoses of sarcoidosis; mycobacterial infections; TSC (definite or possible); cystic lung diseases including genetic diseases; lymphangioleiomyomatosis or diseases associated with lymphatic disorders; history of pneumothorax; pulmonary fibrosis; asthma; histiocytosis X and diabetes mellitus will be included in this protocol. Relatives of patients may also be seen under this protocol. Children with lymphangiomatosis who are two years of age or older may be included. Participants with asthma may be enrolled at Suburban Hospital.

Research volunteers in the pulmonary control group are defined as individuals with no pulmonary disease (e.g. rheumatoid arthritis without evidence of pulmonary disease). Research volunteers in the diabetes control group are defined as individuals with no history of diabetes, coronary artery disease, or pulmonary disease.

Pregnant and or nursing women can be included in accordance with Federal Regulations at Subpart B of 45 CFR 46. Subjects who are pregnant and or nursing will be excluded from procedures during their pregnancy that are greater than minimal risk, until they are no longer pregnant and/or nursing. Procedures that will not be completed while the subject is pregnant and/or nursing including: PFTs, Six Minute Walk Test, thoracentesis, bronchoscopy, and measurements with imaging modalities requiring contrast or with radiation exposure such as Chest x-ray, CT scan, MRI. Allowing subjects to be included in the study may glean important information about individuals with uncommon pulmonary disease during and post pregnancy.

Patients with abnormalities in ADP-ribosyltransferases, ADP-ribosyl-acceptor hydrolases, and their substrates. Children who are two years of age or older may be studied if they have a known defect in ADP-ribosylation, or if they have a family member with a defect in ADP-ribosylation and may be affected.

EXCLUSION CRITERIA:

Exclusion criteria for all participants include:

1. age less than 18 or greater than 90 except for NIH patients with diseases /disorders as described in this protocol (except cystic fibrosis, lymphangiomatosis or defects in ADP-ribosylation) who are 16 years of age or older, patients with cystic fibrosis who are over eight years of age, patients who are two years of age or older with lymphangiomatosis or a known defect in ADP-ribosylation, or who have a family member with a defect in ADP-ribosylation, or unless patient-specific IRB approval is obtained and;
2. inability to obtain reliable pulmonary function testing. As clarification, healthy volunteers, relatives of patients (except as noted for an ADP-ribosylation defect), and asthmatic patients from Suburban Hospital will be excluded if less than 18 or greater than 90 years of age.

Exclusion criteria for participating in the bronchoscopy portion of the study are:

1. presence of any contraindication for fiberoptic bronchoscopy, with lavage and/or bronchial brushing;
2. advanced stage of a pulmonary or a systemic illness such that the risk is judged to be significant even in the absence of a specific contraindication to the procedure
3. allergy to topical anesthetic (e.g., lidocaine)
4. current or recent respiratory infection (within the last 4 weeks)
5. pregnancy or lactation
6. age less than 18 or greater than 65.

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: individuals with pulmonary disease (e.g., alpha 1-antitrypsin deficiency, asthma, chronic obstructive pulmonary disease, cystic fibrosis, sarcoidosis,Wegener s Granulomatosis,Mycobacterium Avium, Tuberous Sclerosis Complex, other cystic lung diseases, lymphangioleiomyomatosis and diseases associated with lymphatic disorders, or history of pneumothorax, history of infection, and genetic mutations consistent with lung pathology)
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 1996-09-13 (Actual)

PRIMARY OUTCOMES:
evaluating the role of hereditary factor | 1 year
  distribution of genetic variants of nitric oxide synthases and other candidate genes involved in pulmonary function

SECONDARY OUTCOMES:
low dose radiation CT scan, and Zoom Scan | on going
  The secondary scan can also be used to obtain a detailed assessment of AML-like tumors and lymphangioleiomyomas in the abdomen or pelvis region when they are detected in the standard chest-abdomen-pelvis CT scan. The enhanced resolution is expected to help classify the tumors without the need for invasive biopsy, for example, by detecting traces of fatty tissue in the tumor to confirm the identity of AML.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
This is a new requirement and the sharing of IPD is not discussed in the protocol.

REFERENCES:
- [Background] Rybicki BA, Beaty TH, Cohen BH. Major genetic mechanisms in pulmonary function. J Clin Epidemiol. 1990;43(7):667-75. doi: 10.1016/0895-4356(90)90037-p. PMID 2370574
- [Background] Welsh MJ, Fick RB. Cystic fibrosis. J Clin Invest. 1987 Dec;80(6):1523-6. doi: 10.1172/JCI113237. No abstract available. PMID 3316277
- [Background] Brantly ML, Paul LD, Miller BH, Falk RT, Wu M, Crystal RG. Clinical features and history of the destructive lung disease associated with alpha-1-antitrypsin deficiency of adults with pulmonary symptoms. Am Rev Respir Dis. 1988 Aug;138(2):327-36. doi: 10.1164/ajrccm/138.2.327. PMID 3264124
- [Derived] Hu-Wang E, Schuzer JL, Rollison S, Leifer ES, Steveson C, Gopalakrishnan V, Yao J, Machado T, Jones AM, Julien-Williams P, Moss J, Chen MY. Chest CT Scan at Radiation Dose of a Posteroanterior and Lateral Chest Radiograph Series: A Proof of Principle in Lymphangioleiomyomatosis. Chest. 2019 Mar;155(3):528-533. doi: 10.1016/j.chest.2018.09.007. Epub 2018 Oct 3. PMID 30291925
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1996-H-0100.html